CLINICAL TRIAL: NCT04790903
Title: A Phase Ib Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Venetoclax in Combination With Polatuzumab Vedotin Plus Rituximab (R) and Cyclophosphamide, Doxorubicin, Prednisone (CHP) in Patients With Untreated BCL-2 Immunohistochemistry (IHC)-Positive Diffuse Large B-Cell Lymphoma
Brief Title: A Study Evaluating the Safety, Efficacy and Pharmacokinetics of Venetoclax in Combination With Polatuzumab Vedotin Plus Rituximab (R) and Cyclophosphamide, Doxorubicin, Prednisone (CHP) in Participants With Untreated BCL-2 Immunohistochemistry (IHC)-Positive Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to discontinue the study based on broader development and strategic prioritisation. The Sponsor concludes there is no benefit-risk impact on the BO42203 study.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BO42203; 2020-002376-12 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — venetoclax; polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venetoclax (Schedule A) (Experimental): Participants enrolled in dosing Schedule A will receive a total of six 21-day cycles of venetoclax treatment for 5 days in combination with Polatuzumab Vedotin + R-CHP (Rituximab, Cyclophosphamide, Doxorubicin and Prednisone) as described below:
  Schedule A: Participants will self-administer Venetoclax orally (PO) once daily (QD) at a dose of 800 mg for 5 consecutive days as follows:
  Cycle 1: 5 consecutive days of dosing on Days 4-8. Cycles 2-6: 5 consecutive days of dosing on Days 1-5.
  Interventions: Drug: Venetoclax; Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone
- Venetoclax (Schedule B) (Experimental): Participants enrolled in dosing Schedule B will receive a total of six 21-day cycles of venetoclax treatment for 10 days in combination with Polatuzumab Vedotin + R-CHP as described below:
  Schedule B: Participants will self-administer Venetoclax orally (PO) once daily (QD) at a dose of 800 mg for 10 consecutive days as follows:
  Cycle 1: 10 consecutive days of dosing on Days 4-10. Cycles 2-6: 10 consecutive days of dosing on Days 1-10.
  Interventions: Drug: Venetoclax; Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Venetoclax — Participants will self-administer Venetoclax, as described in the Arm Descriptions.
Drug: Polatuzumab Vedotin — Participants will receive Polatuzumab Vedotin at a dose of 1.8 mg/kg by intravenous (IV) infusion on Day 1 of Cycles 1-6.
Drug: Rituximab — Participants will receive Rituximab at a dose of 375 mg/m^2 by IV infusion on Day 1 of Cycles 1-6.
Drug: Cyclophosphamide — Participants will receive Cyclophosphamide at a dose of 750 mg/m^2 by IV infusion or bolus on Day 1 of Cycles 1-6.
Drug: Doxorubicin — Participants will receive Doxorubicin at a dose of 50 mg/m^2 by IV infusion or bolus on Day 1 of Cycles 1-6.
Drug: Prednisone — Participants will receive Prednisone orally (PO) at a dose of 100 mg/day on Days 1-5 of Cycles 1-6.

SUMMARY:
This Phase Ib, open-label, multicenter study evaluates the safety, efficacy, and pharmacokinetics of venetoclax in combination with Pola + R-CHP in previously untreated participants with BCL-2 IHC-positive DLBCL. Approximately 50 participants will be enrolled in this study in five consecutive cohorts each consisting of approximately 10 participants.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated participants with CD20-positive DLBCL.
* BCL-2 protein overexpression by IHC, as assessed by local testing.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* International Prognostic Index (IPI) 2-5.
* Life expectancy of more than 6 months.
* Left ventricular ejection fraction (LVEF) ≥ 50%, as determined on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO).
* Availability of archival or freshly collected tumor tissue prior to study enrollment.
* At least one bi-dimensionally fluorodeoxyglucose-avid measurable lymphoma lesion on PET/CT scan, defined as > 1.5 cm in its longest dimension on CT scan.
* Adequate hematopoietic function.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.

Exclusion Criteria:

* Current diagnosis of unclassifiable B-cell lymphoma.
* Prior treatment for indolent lymphoma.
* Current Grade > 1 peripheral neuropathy.
* Prior organ transplantation.
* Prior use of any monoclonal antibody within 3 months and any investigational therapy within 28 days prior to the start of Cycle 1.
* Vaccination with live vaccines within 28 days prior to the start of Cycle 1.
* Prior therapy for DLBCL and High-Grade B-cell Lymphoma (HGBCL) with the exception of palliative, short-term treatment with corticosteroids.
* Recent major surgery (within 6 weeks prior to the start of Day 1 of Cycle 1), other than for diagnosis.
* History of other cancers within 2 years prior to screening.
* Any active infection that, in the opinion of the investigator, would impact participant safety within 7 days prior to Day 1 of Cycle 1.
* Serious infection requiring oral or IV antibiotics within 4 weeks prior to Day 1 of Cycle 1.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study.
* Positive test for Hepatitis B/C Viruses (HBV/HCV) and Human T-cell Leukemia Virus (HTLV)-1.
* Known infection with HIV.
* History of progressive multifocal leukoencephalopathy.
* Suspected active or latent tuberculosis.
* Clinically significant history of liver disease, including viral or other hepatitis or cirrhosis.
* Substance abuse, including non-prescription drug and alcohol dependence, within 12 months prior to screening.
* Pregnant or breastfeeding, or intending to become pregnant during the study within 6 months after the final dose of venetoclax, 9 months after the final dose of polatuzumab vedotin, or 12 months after the final dose of rituximab.
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion.
* Malabsorption syndrome or other condition that would interfere with enteral absorption.
* Blood transfusion within 14 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Cycle 1 Day 1 up to but not including Cycle 3 Day 1 (Cycle length = 21 days)

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 4 years
Complete Response (CR) rate at the end of treatment | Up to 4 years
  Assessed by the investigator on PET and computed tomography (PET/CT) scans according to the Lugano Response Criteria for Malignant Lymphoma (Cheson et al. 2014)
Objective Response Rate (ORR) at the end of treatment | Up to 4 years
  Defined as the proportion of patients with a CR or a partial response (PR), as determined by the investigator on PET/CT scans according to the Lugano 2014 Response Criteria
Duration of Response (DOR) | Up to 4 years
  Defined as the time from the first occurrence of a documented objective response (a PR or a CR) to disease progression, relapse, or death from any cause (whichever occurs first), as determined by the investigator according to the Lugano 2014 Response Criteria
Progression-Free Survival (PFS) | Up to 4 years
  Defined as the time from the date of first study treatment to the first occurrence of disease progression or relapse, as assessed by the investigator, according to the Lugano 2014 Response Criteria, or death from any cause, whichever occurs earlier
Plasma Concentrations of Venetoclax at specified timepoints | Up to 4 years
Plasma Concentrations of Polatuzumab Vedotin analytes at specified timepoints | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- United States (3):
  - NYU Langone Hospitals, NYU Langone Rusk Ambulatory Surgical Pharmacy, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SARAH CANNON RESEARCH INST.; Tennessee Oncology, PLLC, Nashville, Tennessee
- France (7):
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - CHU Montpellier - Saint ELOI, Montpellier
  - CHU de Nantes; Cancéro-dermatologie, Nantes
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud; Service d'Oncologie Médicale, Pierre-Bénite
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
- Italy (5):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale;s.c. Ematologia Oncologica, Napoli, Campania
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola Malpighi; Dip. Scienze Mediche e Chirurgiche, Bologna, Emilia-Romagna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST; Farmacia Oncologica, Meldola, Emilia-Romagna
  - Ospedale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Pisana-Ospedale Santa Chia, Pisa, Piedmont
- Spain (5):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital de la Santa Creu i Sant Pau; Servicio de Dermatologia, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Univ. Gregorio Maranon, Madrid
  - Hospital Universitario La Fe; Servicio de Farmacia, Valencia

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).